CLINICAL TRIAL: NCT06774833
Title: Effect of Self-initiated Perturbation-based Balance Training on the Postural Stability of Community-dwelling Older Adults with an Increased Risk of Falling: a Randomized Controlled Trial
Brief Title: Self-initiated Perturbation-based Training in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20240505001
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Healthy Subjects (HS)
Keywords: Perturbation; Step training; Falls

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to SePBT or conventional balance training group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-initiated perturbation-based balance training group (Experimental): This group will receive two sessions of self-initiated perturbation-based balance training.
  Interventions: Behavioral: Self-initiated perturbation-based balance training
- Conventional balance training group (Active Comparator): This group will receive two sessions of balance and strength training.
  Interventions: Behavioral: Conventional balance training

INTERVENTIONS:
Behavioral: Self-initiated perturbation-based balance training — This group will receive two 30-minute training sessions over two weeks, with one session per week. Participants will be required to recover their balance upon self-initiated perturbation.
  Arms: Self-initiated perturbation-based balance training group
Behavioral: Conventional balance training — This group will receive two 30-minute training sessions over two weeks, with one session per week. Participants will be instructed to perform balance and strength training. The same training duration and format will be used as the Self-initiated perturbation-based balance training group.
  Arms: Conventional balance training group

SUMMARY:
This is a single-blinded study. Participants will be randomly assigned to self-initiated perturbation-based balance training (SePBT) group or control (conventional balance training) group. Kinematic and Kinetic changes following SePBT group compared to control will be investigated.

DETAILED DESCRIPTION:
Participants will be randomly assigned to two groups receiving SePBT or control group. All participants will give their written informed consent before baseline assessment. The study will be reported and conducted in line with the CONSORT statement. Participants will be recruited via convenient sampling in the local community. After baseline assessment, both groups will go through two 30-minute training session over two weeks. Between-group differences in behavior will be examined before and after training to identify training-induced changes in postural stability. Retention of the changes in the postural stability will be assessed four months after the training period. Incidents of falls will be followed up for 12 months after training.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged 60 years old or older
* Able to communicate effectively in Cantonese or Mandarin
* Able to walk independently on level ground for at least 30 minutes
* Abbreviated Mental Test (Hong Kong version) scores≥6
* Have fallen in the preceding year, have concerns about falling, or feel unsteady while walking or standing.

Exclusion Criteria:

* Uncorrected vision or hearing impairment
* Osteoporosis
* Hip or knee replacement within the last year
* Have musculoskeletal, cardiovascular, mental, or neurological disorders that preclude their participation in the assessment or intervention safety

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postural stability | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Postural stability at the recovery steps after the perturbation will be calculated as the distance between the absolute center of mass (CoM) position in an anteroposterior direction relative to the closest edge of the Base of Support (BoS) normalized by foot length. The absolute CoM position and BoS position will be traced by the motion capture system synchronized with the force plates embedded underneath the slip-treadmill belts.

SECONDARY OUTCOMES:
Generic balance ability | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Generic balance ability will be assessed by the Mini-BESTest. It contains 8 test items and each item will score between 0 and 3 and the total scores will range from 0 to 24, with higher scores denoting better balance ability.
Mobility | Pre-intervention, 1 week after intervention and 4 months after intervention
  Mobility will be assessed by Timed Up and Go test (in the unit of seconds).
Number of real-life falls | 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 7 months, 8 months, 9 months, 10 months, 11 months, and 12 months after the intervention.
  The number of real-life falls in months after randomization will be recorded. Fall circumstances and related injuries will be required via phone contact. A fall is defined as an event resulting in a person unintentionally coming to rest on the ground or other lower level, not as the result of a major intrinsic event (e.g., syncope, stroke, or overwhelming hazard such as an earthquake).
Responsive postural adjustment upon translation | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Responsive postural adjustment upon translation will be assessed through Motor Control Test and Adaptation Test on a computerized dynamic posturography (Bertec® Balance Advantage® Dynamic system, Bertec® Corporation, Columbus, USA). During the Motor Control Test, participants will be requested to maintain their standing balance in response to 12 translations of the standing platform in either forward or backward direction with medium and large amplitudes. Weight symmetry, latency of reaction and amplitude of sway will be recorded. Full-body safety harness will be worn throughout the tests to protect the participants from any potential loss of balance.
Responsive postural adjustment upon tilting | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Responsive postural adjustment upon tilting will be assessed through Adaptation Test on a computerized dynamic posturography (Bertec® Balance Advantage® Dynamic system, Bertec® Corporation, Columbus, USA). During the Adaptation Test, the force platform will either tilt up or down for a total of 10 repetitions. Sway energy will be recorded. Full-body safety harness will be worn throughout the tests to protect the participants from any potential loss of balance.
Dynamic balance | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Dynamic balance will be assessed by Alternative Step Test (in the unit of seconds).
Balance confidence | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Balance confidence will be measured with the Chinese version of the shortened version of Activities-specific Balance Confidence Scale (ABC-6). The scale value is from 0 to 100, with higher values representing higher balance confidence.
Functional lower body strength | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Functional lower body strength will be assessed by Five-time Sit to Stand Test (in the unit of seconds).
Cognitive flexibility and executive function | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Cognitive flexibility and executive function will be assessed by Trial Making Tests A and B (in the unit of seconds).
Number of laboratory falls | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Participants will be exposed to one trip-like perturbation and slip-like perturbation on each foot at an unexpected time. The number of falls upon perturbations will be recorded.
Cognitive impairment | Pre-intervention.
  Cognitive impairment will be assessed by Abbreviated Mental Test (AMT). AMT is a 10-item test, with a 10-point scale. A score less than 6 suggests a significant cognitive deficit.
Depressive symptoms | Pre-intervention.
  Depressive symptoms will be assessed by Five-Item Geriatric Depression Scale. Participants will be asked to answer 5 questions as yes or no. The answer "no" for the first question and "yes" for the other four questions will be evaluated for depression.
Personality traits | Pre-intervention.
  Personality traits assessed by Ten-Item Personality Inventory. It has 10 items, each item adopts a 5-level score of 1 (Disagree strongly) to 5 (Agree strongly), and a higher dimension score indicates a stronger individual's personality proneness.
Generic preference-based quality-of-life | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Generic preference-based quality-of-life will be assessed by five-level EuroQol five-dimensional questionnaire (EQ-5D-5L). The EQ-5D-5L essentially consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  In the EQ-5D descriptive system, each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Each health state is identified by a five-digit code, with 11111 representing the best and 55555 the worst possible health state.
  In the EQ CAS, the scale value is from 0 to 100, with higher values representing higher balance confidence.
Muscle activations | Pre-intervention, 1 week after intervention and 4 months after intervention.
  Muscle activations will be assessed by surface electromyography using an electromyography system (Trigno IM, Delsys Inc., Natick, MA, USA). Fourteen electrodes are placed bilaterally over erector spinae, rectus abdominis, gastrocnemius medialis, biceps femoris, rectus femoris, tibialis anterior, and gluteus medius according to the SENIAM guidelines (www.seniam.org) by the physical therapist.
Physical activity | Pre-intervention, and 4 months after intervention
  Physical activity will be assessed by the Physical Activity Scale for the Elderly. This questionnaire will ask participants to recall their activity over the last 7-days. Activity types include sitting, walking, sport/recreation, exercise, occupational and household. A total score for physical activity can be calculated using these answers and the predetermined weights associated with each activity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No